CLINICAL TRIAL: NCT07057960
Title: Group Social Work Intervention in Improving Peer Relationships of Children in Institutional Care: A Mixed Methods Study
Brief Title: Group Social Work Intervention in Improving Peer Relationships
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Rabia Ruveyda Yigit, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/564
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Bullying
Keywords: Peer Relationships; Peer Bullying; Cognitive Behavioral Therapy; Children; Institutionalized; Group Social Work Intervention
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Social Work Intervention Based on CBT (Experimental): The experimental group will participate in a group intervention based on cognitive behavioral therapy (CBT). The sessions will be conducted by the researcher twice a week over a period of five weeks.
  Interventions: Other: Group Social Work Intervention Based on Cognitive Behavioral Therapy
- Wait-List Control Group (Other): The control group will consist of children placed on a waiting list. These children will not receive any intervention while the experimental group is undergoing the program. Following the completion of the intervention for the experimental group and the collection of post-test data, the same intervention will be offered to the children in the control group.
  Interventions: Other: Group Social Work Intervention Based on Cognitive Behavioral Therapy

INTERVENTIONS:
Other: Group Social Work Intervention Based on Cognitive Behavioral Therapy — The aim of the intervention is to modify children's bullying-related cognitions and enhance peer relationships through cognitive restructuring, achieved by increasing awareness of cognitions, emotions, and behaviors among children in institutional care.
  The content of the intervention was developed using the core principles and techniques of cognitive behavioral therapy.

SUMMARY:
The aim of this mixed-methods study is to examine the effect of a group social work intervention, based on cognitive behavioral therapy, on bullying-related cognitions and peer relationships among boys in institutional care. Additionally, the study will explore the experiences and perspectives of participants in the experimental group regarding the intervention.

DETAILED DESCRIPTION:
In this study, designed as a mixed-methods research, a mixed-methods experimental (or intervention) design will be employed, in which participants' experiences and opinions about the intervention are embedded within an experimental framework.

In the first phase, quantitative data will be collected and analyzed to assess the effectiveness of a group social work intervention on peer relationships and bullying-related cognitions among boys in institutional care. In the linkage phase, findings from the quantitative analysis will inform the selection of qualitative research participants and the development of the interview protocol. Subsequently, qualitative data will be gathered and analyzed to gain deeper insight into the experiences of the experimental group participants regarding the intervention, and to enhance the interpretation of the quantitative findings. Finally, the results from both data types will be integrated and interpreted.

The quantitative component of the study will be conducted as a parallel-group, single-blind, randomized, waiting list-controlled experimental design. After being informed about the study, all participants who provide written informed consent will be screened for eligibility. Those who meet the inclusion criteria will be randomly assigned, in a 1:1 ratio, to either the experimental group or the waiting list control group. The implementation phase of the quantitative study will consist of a group social work intervention.

The qualitative component of the study is designed as a phenomenological research approach. In-depth interviews will be conducted to explore the experiences of participants in the experimental group regarding the intervention, as well as their views on its content, applicability, and perceived effects. These interviews also aim to provide a deeper understanding of the quantitative findings. A semi-structured interview guide, to be developed during the linkage phase, will be used to collect the qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 18 years
* Residing in institutional care for at least three months
* Literate
* Voluntarily agree to take part in the research

Exclusion Criteria:

* Diagnosis of an acute psychotic disorder
* Previous participation in a similar intervention based on cognitive behavioral therapy
* Missing at least two intervention sessions (after study initiation)
* Leaving the institution or being transferred to another institution during the course of the study (after study initiation)
* Withdrawal of informed consent (after study initiation)

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Peer Relationship Scale | T0 (Pre-test) T1 (15 days after the end of the procedure)
  The scale was developed to assess adolescents' peer relationships. It comprises 29 items across four sub-dimensions: Intimacy, Popularity, Trust, and Insightfulness. The items are rated on a 5-point Likert scale ranging from 1 (Strongly disagree) to 5 (Completely agree.). The total possible score on the scale ranges from 29 to 145, with higher scores indicating more positive peer relationships.
Inventory of Cognitions Related to Bullying for Children | T0 (Pre-test) T1 (15 days after the end of the procedure)
  The scale was developed to assess cognitive characteristics associated with peer bullying in children. It consists of 22 items rated on a 4-point Likert scale, ranging from 1 (Not true at all) to 4 (Completely true). The total score on the scale ranges from 22 to 88. Higher scores indicate stronger cognitive acceptance of bullying, suggesting that bullying is perceived as more normal and acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Feyzal Kesen, Study Director — Selcuk University
Locations (1):
- Karatay Çocuk Evleri Sitesi Müdürlüğü, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gökkaya, F., ve Tekinsav-Sütçü, S. (2015). Çocuklar için Zorbalıkla İlgili Bilişler Ölçeğinin geliştirilmesi ve psikometrik özelliklerin değerlendirilmesi. Anadolu Psikiyetri Dergisi, 16(Ek sayı-1), 54-63.
- [Background] Aydogdu F. Developing a Peer Relationship Scale for Adolescents: a validity and reliability study. Curr Issues Personal Psychol. 2021 Oct 14;10(2):164-176. doi: 10.5114/cipp.2021.109461. eCollection 2022. PMID 38013922